CLINICAL TRIAL: NCT05796973
Title: Syöpäpotilaan Ennusteen Parantaminen Muuttamalla syövän mikroympäristöä ja Metaboliaa Liikunnalla ja lääkkeellisesti - Measuring Oncological Value of Exercise and Statin
Brief Title: Measuring Oncological Value of Exercise and Statin
Acronym: MOVES
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); Aalto University (Other); University of Helsinki (Other); University of Turku (Other)
Responsible Party: Principal Investigator, Teemu Murtola, Professor of Urology, Chief Physician, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-001982-34
Record Dates: First submitted 2023-02-13; First posted 2023-04-04 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer; Breast Cancer; Kidney Cancer; Ovarian Cancer; Metastatic Breast Cancer; Metastatic Kidney Cancer; Metastatic Renal Cell Carcinoma; Metastatic Renal Cancer; Metastatic Prostate Cancer; Metastatic Prostate Adenocarcinoma; Metastatic Ovarian Cancer; Metastatic Ovary Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Kidney Neoplasms; Ovarian Neoplasms; Carcinoma, Renal Cell | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: The patients are randomized equally into three groups: 1/3 into guided exercise group, 1/3 into guided exercise and statin-treatment group and 1/3 into non-guided exercise group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Guided physical exercise arm (Experimental): 20 patients from each type of cancer (altogether 80) are randomized to a 3 months guided physical exercise arm. At the beginning of the intervention the patients' physical condition and body composition are measured. After that an exercise program begins. All subjects participate in physical exercise program twice a week for three months. At the end of the intervention, the physical condition and body composition are measured again. During the follow-up after the intervention the patients are advised to exercise regularly. Physical condition and body composition are measured again after 6 months. Exercise activity is asked during each follow-up visit.
  In addition, as a separate group, 20 patients from each type of cancer (altogether 80) who are already using statin medication are randomized to this arm.
  Interventions: Behavioral: Guided physical exercise
- Atorvastatin arm (Experimental): 20 patients from each type of cancer (altogether 80) are randomized to a 3 months guided physical exercise + atorvastatin (40 mg QD) arm. At the beginning of the intervention the patients' physical condition and body composition are measured. After that an exercise program begins. All subjects participate in physical exercise program twice a week for three months. At the end of the intervention, the physical condition and body composition are measured again. During the follow-up after the intervention the patients are advised to exercise regularly. Physical condition and body composition are measured again after 6 months. Exercise activity is asked during each follow-up visit.
  Interventions: Behavioral: Guided physical exercise; Drug: Atorvastatin
- Non-guided physical exercise arm (Active Comparator): 20 patients from each type of cancer (altogether 80) are randomized to a non-guided physical exercise arm. The patients' physical condition and body composition are measured at baseline. The control group is advised of the benefits of physical exercise and they get an exercise program to follow. Participants in the control group exercise on their own. The physical condition and body composition of this group is also measured at three months and six months after baseline to detect changes. After that the patients are given advise to exercise regularly and this is asked during each follow-up visit.
  In addition, as a separate group, 20 patients from each type of cancer (altogether 80) who are already using statin medication are randomized to this arm.
  Interventions: Other: Independent exercise

INTERVENTIONS:
Behavioral: Guided physical exercise — Patients will be participating in guided physical exercise program regularly two times / week at a sports facility and guided by a professional trainer. They will participate in aerobic and resistance exercises during the sessions.
  Arms: Atorvastatin arm; Guided physical exercise arm
Drug: Atorvastatin — Patients will be participating in guided physical exercise program regularly two times / week at a sports facility and guided by a professional trainer. They will participate in aerobic and resistance exercises during the sessions. In addition to the exercise program they will be given atorvastatin 40 mg QD medication.
  Arms: Atorvastatin arm
Other: Independent exercise — The control group is advised of the benefits of physical exercise and they get an exercise program to follow. Participants in the control group exercise on their own.
  Arms: Non-guided physical exercise arm

SUMMARY:
The aim of the study is to find out whether supervised physical exercise during cancer drug treatment improves the effectiveness of the treatment in metastasized breast, kidney, ovarian and prostate cancer compared to unsupervised exercise. In addition, the investigators are investigating whether the use of atorvastatin combined with guided group exercise training would further improve the response to cancer treatment.

DETAILED DESCRIPTION:
Despite the marked differences between different malignancies' genetic, metabolic, and prognostic factors, hypoxia and adaptation of metabolic changes favoring hypoxic microenvironment are common factors in most solid tumors. Hypoxic microenvironment provides cancer cells multiple advantages: protection from immune system, somatic mutations leading to more aggressive form of cancer, and cancer cells that are adjusted to hypoxic conditions are more prone to form metastases. One possible mechanism for cancer cell to adjust to hypoxic microenvironment is related to lipid metabolism; lipids are known to accumulate into cancer cells in many cancer types. One of the most promising ways to reduce hypoxia in solid tumors is to increase physical exercise. Furthermore, tumors' lipid metabolism can be affected by treatment with cholesterol-lowering statins, which decreases serum cholesterol levels and inhibits cancer cells' own lipid synthesis.

The aim of this randomized clinical trial is to investigate if supervised group exercise will improve response to cancer drug treatment in metastasized breast, kidney, prostate, and ovarian cancer compared to unsupervised exercise. The investigators will also evaluate if atorvastatin treatment in combination with guided group exercise can promote even better treatment responses than exercise alone. Exercise program includes aerobic and resistance training.

This study is a randomized phase III study testing the research hypothesis for the first time in humans. A total of 240 cancer patients (n=60/cancer type) will be recruited into the study and randomized 1:1:1 into three different groups, i.e. 20 people in each group from each cancer type:

1. 3 months of supervised group exercise
2. 3 months of supervised group exercise and at the same time atorvastatin 40 mg/day
3. to a control group that exercises voluntarily without guidance.

In addition, as a separate group, a total of 160 cancer patients (40/cancer type) who are already using statin medication will be recruited for the study and randomized 1:1 into two groups: 1) 3 months of supervised group exercise and 2) independent exercise (a control group that exercises voluntarily without guidance).

Before the study begins, the patients are informed orally and in writing about the study. The patients who agree to participate in the study sign an informed consent.

The patient follow-up time in each group is two years in 3 months intervals (first visit and 8 follow-up visits) in conjunction with standard cancer treatment follow-up visits. Blood and urine samples and questionnaire data are collected at baseline and at each follow-up visit. Body composition and physical performance are measured at baseline and twice after the intervention. Patients QoL and experiences of exercise are measured in qualitative interviews (in the group participating the qualitative sub-study).

The main response variables are

1. cancer progression during cancer treatment based on imaging, symptoms or laboratory findings and
2. mortality of the patients.

   The other variables of interest in this study are:
3. Hypoxia markers
4. Tolerability of treatment
5. Body composition
6. Physical performance
7. The extent of hypoxia, as measured by PET scans, in participants of the sub-study

4) Quality of life, perceived pain, depressive symptoms, nutrition and relationships.

Adverse events from cancer treatment and treatment interruptions are also monitored.

ELIGIBILITY:
Inclusion Criteria:

* The patient has metastatic prostate cancer, breast cancer, ovarian cancer or kidney cancer confirmed histologically and by imaging, for which 1st-line cancer drug treatment is started
* Prostate cancer: First course of docetaxel treatment or second-generation antiandrogen treatment for metastatic prostate cancer.
* Breast cancer: First-line medical treatment of metastatic breast cancer regardless of hormone receptor status.
* Kidney cancer: Kidney cancer, for which 1st-line cancer drug treatment is started as tki monotherapy and/or IO monotherapy or as a combination therapy.
* Ovarian cancer: stage III or IV cancer for which chemotherapy treatment is started.
* The patient agrees to the study and signs a written informed consent.
* Adult (18 years=>) women (breast, ovarian and kidney cancer) and men (prostate and kidney cancer) are recruited for the study.
* In women, the use of a reliable contraceptive during the intervention

Exclusion Criteria:

* High risk of bone fractures
* Inability to physical exertion and/or unsuitability for cancer drug treatment
* Poor co-operation ability for psychological reasons
* Active use of cholesterol-lowering drugs
* Severe liver or kidney failure
* Troublesome side effects that occurred in the past during cholesterol medication
* Continuous use of medicinal substances that interact with atorvastatin during the study period
* A special group of subjects according to the EU Clinical Trials Regulation 536/2014 (e.g. pregnant or lactating women)

Exclusion criteria in patients who are already using statin medication before the study:

* High risk of bone fractures
* Inability to physical exertion and/or unsuitability for cancer drug treatment
* Poor co-operation ability for psychological reasons
* Severe liver or kidney failure
* A special group of subjects according to the EU Clinical Trials Regulation 536/2014 (e.g. pregnant or lactating women)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to cancer progression | From randomization until the date of first documented progression, assessed at twelve week intervals up to 24 months
  Radiological progression • Radiological progression of the disease according to RECIST criteria (version 1.1.) compared to the situation at the start of cancer treatment in all cancer types. If the cancer treatment includes the use of immune checkpoint inhibitors, the imRECIST criteria are applied to evaluate the response
  In addition, the disease is considered advanced if both of the criteria below are met:
  * Biochemical progression:
    * PSA progression in prostate cancer, (three consecutive PSA increases measured at least one week apart, two > 50% increases from the lowest PSA level and PSA > 2 ng/ml) with testosterone at castration level (< 50 ng/ml or 1.7 nmol/l)
    * Ca15-3 marker increase in breast cancer (three consecutive marker increases that the clinician considers significant)
    * In ovarian cancer, ca12-5 marker increase (three consecutive marker increases that the clinician considers significant)
  * Clinical progression o ECOG 3 or less (long-term)
Mortality | From randomization until the date of death, assessed up to 24 months
  Time to death from the beginning of the first-line medication

SECONDARY OUTCOMES:
Hypoxia markers in serum (VEGF, HIF1-alpha, carboanhydrase IX, LADH) | At baseline and at 3 months
  Hypoxia markers in the serum
Tolerability of treatment | From date of randomization, assessed at twelve week intervals up to 24 months
  Incidence of grade 3 or worse adverse events during cancer treatment
Fat/muscle ratio as measured with impedance test | At baseline and at 3 and 6 months
  Body composition measurement before and after the intervention
Physical performance with standardized muscle strength tests | At baseline and at 3 and 6 months
  Muscle strength tested with three standardized tests (squat test, core dynamic strength test, biceps flexion test) before and after the intervention.
Changes in tissue hypoxia | At baseline and at 3 months
  The amount of hypoxia in cancer foci determined by PET-CT scan using specific hypoxia-sensitive tracers in a sub-study
Changes in quality of life | At baseline and at 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months and 24 months
  EORTC-QLQ-C30 questionnaire to measure quality of life, score from 0 to 100. A high scale score for a functional scale represents a higher level of functioning, a high score for a symptom scale represents higher level of symptoms.
Depressive symptoms | At baseline and at 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months and 24 months
  Patient Health Questionnaire (PHQ-9), score from 0 (no depression) to 27 (severe depression).
Severity of pain | At baseline and at 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months and 24 months
  The severity of pain and its impact on functioning. Brief Pain Inventory questionnaire including 9 items. Pain severity scale from 0 (no pain) to 10 (worst pain), pain interference from 0 (does not interfere) to 10 (completely interferes).
Nutritional status | At baseline and at 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months and 24 months
  Mini Nutritional Assessment (MNA) questionnaire. A score of 7 or less (malnutrition) to 24-30 (normal nutrition).
Relationship satisfaction | At baseline and at three months, twelve months and 24 moths.
  The relationship questionnaire consists of two previously used, validated measures: Dyadic Adjustment Scale (DAS) and Marital Communication Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Teemu Murtola, MD PhD Prof, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Länsi-Suomi, Finland

IPD SHARING:
Plan to Share IPD: No